CLINICAL TRIAL: NCT03578302
Title: The Heidelberg Engineering BI US Evaluation Study
Status: Completed | Type: Observational
Sponsor: Heidelberg Engineering GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: B-2018-1
Record Dates: First submitted 2018-06-21; First posted 2018-07-06 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2019-01

CONDITIONS: Normal Eyes; Eye Abnormalities
MeSH Terms: conditions — Eye Abnormalities

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Anterior Segment Pathology: single measurement Anterior Segment Pathology
  Interventions: Device: BI Anterior Segment Mode
- All except Anterior Segment Pathology: 3 repeat measurements with and without dilation for all eyes except Anterior Segment Pathology
  Interventions: Device: BI Anterior Segment and IOL Biometry Mode

INTERVENTIONS:
Device: BI Anterior Segment Mode — Single eye measurement in Anterior Segment Mode
  Groups: Anterior Segment Pathology
Device: BI Anterior Segment and IOL Biometry Mode — Eye measurement 3 times with and without dilation in IOL biometry and Anterior Segment mode
  Groups: All except Anterior Segment Pathology

SUMMARY:
Evaluation of defined parameters measured in pathological and non-pathological eyes with the Heidelberg BI

DETAILED DESCRIPTION:
The primary objectives of this study are to assess the feasibility to acquire acceptable images and to assess repeatability

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Able and willing to undergo the test procedures, sign informed consent, and follow instructions

   At least one of the following:
3. Eyes with Normal Anterior Segment
4. Eyes with Cataract
5. Eyes without a Crystalline Lens
6. Eyes with Corneal Abnormality
7. Eyes with Anterior Segment Pathology

Exclusion Criteria:

1. Subjects unable to read or write
2. Active infection or inflammation in one or both eyes
3. Insufficient tear film or corneal reflex
4. Physical inability to be properly positioned at the study devices or eye exam equipment
5. Inability to fixate
6. Rigid contact lens wear during past 2 weeks
7. Soft lenses, in the study eye, if worn, should be removed at least one hour prior to the measurements *Note: Eyes with risk for acute angle closure glaucoma are excluded from the dilated portion of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with:
  1. Eyes with Normal Anterior Segment or
  2. Eyes with Abnormal Anterior Segment, including Eyes with Cataract Eyes without a Crystalline Lens Eyes with Corneal Abnormality Eyes with Anterior Segment Pathology
Sampling Method: Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2018-05-22 (Actual); Primary Completion 2018-12-03 (Actual); Study Completion 2018-12-03 (Actual)

PRIMARY OUTCOMES:
Percentage of successfully scanned biometry images of the eye | 1 day
  Percentage of successfully scanned biometry images of the eyes per scan mode. Success is defined as agreement of the subjective assessment of the operator and the auto assessment of the device.
Repeatabiltiy of specific parameters of the biometry images of the eye | 1 day
  Repeatability of specific parameters stratified by different eye pathologies

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Dul, OD, Principal Investigator — State University of New York College of Optometry
Locations (1):
- State University of New York College of Optometry, New York, New York, United States